CLINICAL TRIAL: NCT05080816
Title: Effects of Parenteral and Enteral Nutrition on Skeletal Muscle Genomics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: MB3
Record Dates: First submitted 2021-06-10; First posted 2021-10-18 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Muscle Loss
Keywords: Skeletal muscle
MeSH Terms: conditions — Muscular Atrophy | interventions — Parenteral Nutrition; Parenteral Nutrition, Total; Enteral Nutrition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Persons responsible for genomic/transcriptomic/proteomics analyses are blinded. All samples are coded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Parenteral nutrition (Active Comparator): Overnight infusion of parenteral nutrition. Supplied as all-in-one-bag format. Infusion rate of 0.2 g N/kg/day.
  Interventions: Dietary Supplement: Parenteral nutrition (PN)
- Enteral nutrition (Active Comparator): Oral nutrition drink. 2 * 200 ml on the night before operation. 1* 200 ml on the morning of operation day.
  Interventions: Dietary Supplement: Enteral nutrition
- control (Placebo Comparator): Overnight infusion of crystalloid fluid (Ringer acetate) infused at the same rate (ml/kg) as intervention PN
  Interventions: Other: Control

INTERVENTIONS:
Dietary Supplement: Parenteral nutrition (PN) — Overnight infusion of parenteral nutrition. Supplied as all-in-one-bag format. Infusion rate of 0.2 g N/kg/day.
  Other Names: Total parenteral nutrition (TPN)
  Arms: Parenteral nutrition
Dietary Supplement: Enteral nutrition — Oral nutrition drink. 2 * 200 ml on the night before operation. 1* 200 ml on the morning of operation day.
  Other Names: nutrition drink
  Arms: Enteral nutrition
Other: Control — Overnight infusion of crystalloid fluid (Ringer acetate) infused at the same rate (ml/kg) as intervention PN
  Arms: control

SUMMARY:
The study investigates effects related to muscle protein metabolism at provision of Parenteral or enteral nutrition

DETAILED DESCRIPTION:
Randomized study investigation alterations in muscle protein metabolism at provision of parenteral or enteral (oral drink) nutrition. The study uses a genomic/transcriptomic/proteomic approach to evaluate factors related to activation of skeletal muscle protein synthesis and protein degradation. Patients scheduled for major gastrointestinal surgery are included. Muscle specimens are collected during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Major gastrointestinal surgery.
* Assumed need of post-operative nutrition support.

Exclusion Criteria:

* Insulin dependent diabetes.
* Steroid medication.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2018-10-18 (Actual)

PRIMARY OUTCOMES:
Muscle protein metabolism | ~12-14 hours.
  Alterations in skeletal muscle gene expression quantified by microarray

CONTACTS AND LOCATIONS:
Overall Officials: Britt-Marie Iresjö, Ph.D, Principal Investigator — Göteborg University
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Region Västra Götaland, Sweden

REFERENCES:
- [Derived] Iresjo BM, Smedh U, Engstrom C, Persson J, Martensson C, Lundholm K. A randomized translational study on protein- and glucose metabolism in skeletal muscles evaluated by gene-ontology, following preoperative oral carbohydrate loading compared to overnight peripheral parenteral nutrition (PPN) before major cancer surgery. J Transl Med. 2024 Jul 22;22(1):675. doi: 10.1186/s12967-024-05484-1. PMID 39039509